CLINICAL TRIAL: NCT04938739
Title: Effect of Cognitive Behavioral Therapy in Patients With Chronic Nonspecific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Manar Abd El galil Aneis, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Manis_MSc
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Low Back Pain, Mechanical
MeSH Terms: conditions — Low Back Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral therapy (Experimental): to modify any erroneous beliefs about pain and disability and to promote coping strategies and self-efficacy through a graded activity.
  Interventions: Other: Cognitive Behavioral Therapy; Other: Home program exercises
- Home program exercises (Active Comparator): Patients in both groups carried out exercise therapy for six weeks. There will be an educational session for each patient to make sure the exercises will be done successfully and supervision once per week.
  Interventions: Other: Home program exercises

INTERVENTIONS:
Other: Cognitive Behavioral Therapy — The first 6 sessions: the cognitive part was explained with the support of a PowerPoint presentation using diagrams, images, and texts. The therapist explained the lumbar engine behavior, the neurophysiologic basis of pain, the importance of the participant's involvement in the treatment (e.g., coping and motivation), and the maintenance of good ergonomics which was aimed at modifying the physiologic response to the pain system.
  The second 12 sessions: concepts viewed in the first session were revised; as well, the operant and respondent parts were explained.
  Arms: Cognitive Behavioral therapy
Other: Home program exercises — Each session will include 10 minutes of aerobic activity (walking or stationary bicycle), followed by five types of muscle stretches and eight types of ground exercises aimed at strengthening the lumbar muscles responsible for stabilization.

SUMMARY:
The purpose of the study is to determine the effectiveness of cognitive-behavioral therapy on functional outcomes, pain, and pain-related anxiety in patients with chronic nonspecific low back pain

DETAILED DESCRIPTION:
Back pain has considerable negative effects on the quality of life of affected individuals. Individuals with new-onset back pain have an increased risk of lower quality of life scores, and the negative effect on quality of life increases with persistent pain. Patients with chronic back pain report a quality of life that is lower than individuals without pain and that is comparable to those of individuals with life-threatening diagnoses. In addition, back pain is associated with worry and fears, particularly about the (sense of) self and socialrelationships and especially when pain persists longer than expected.

ELIGIBILITY:
Inclusion Criteria:

1. Thirty patients with non-specific chronic low back pain from both sexes will be included.
2. Subjects with normal body mass index (18 to 25).
3. The age of patients range from 20 to 35 years.
4. Duration of pain more than 3 months up to 2 years.
5. Normal cognition score 26 or above according to MoCA Scale.7. Highly educated at least high school.

Exclusion Criteria:

The patients will be excluded if they have any of the followings:

1. Lumbar canal stenosis.
2. Lumbar discogenic lesions.
3. Any inflammatory arthritis, tumors, infection involving the lumbar spine.
4. Patients with decreased range of motion secondary to congenital anomalies, muscular contracture or bony block.
5. Previous lumbar surgery or trauma.
6. Subjects with a history of any neurologic disease.
7. Cauda equina Syndrome.
8. Patients suffering from psychological, cognitive or emotional disturbance.
9. Patients who had previously participated in cognitive behavioral therapy.
10. Deafness and blindness.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Assessing the change in pain intensity | Baseline and 6 weeks post-intervention
  Assessment via using visual analogue scale A tool used to help a person rate the intensity of certain sensations and feelings, such as pain. The visual analog scale for pain is a straight line with one
Assessing the change in back function | Baseline and 6 weeks post-intervention
  Assessment via using Oswestry Low Back Pain Disability Index It is a 10-item self assessing questionnaire; each item contains 6 levels of answers that can be scored from 0 to 5.

SECONDARY OUTCOMES:
Assessing the change in anxiety related to pain | Baseline and 6 weeks post-intervention
  Assessment via using pain anxiety symptom scale (PASS) is a 20-item self-report scale that measures components of pain-related anxiety, including cognitive anxiety, escape and avoidance, fearful appraisals of pain, and physiological anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Manar Abdelgalil, Abdelgalil, Principal Investigator — Horus University in Egypt
Locations (1):
- Outpatient clinic - Faculty of Physical Therapy - Cairo University, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No